CLINICAL TRIAL: NCT04289090
Title: Sevoflurane Versus Propofol on Optic Nerve Sheath Diameter During Anesthesia in Steep Trendelenburg Position
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1281970-5
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Percentage of Change in ONSD During Anesthesia With Sevoflurane Versus Propofol in Two Groups of Patients
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Group A will begin anesthesia maintenance with sevoflurane-only, then will be switched after 30 minutes to anesthesia with propofol-only. Group B will begin anesthesia with propofol-only then will be switched to sevoflurane-only.
Who Masked: Participant
Masking Description: Group A will begin anesthesia maintenance with sevoflurane-only, then will be switched after 30 minutes to anesthesia with propofol-only. Group B will begin anesthesia with propofol-only then will be switched to sevoflurane-only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will begin anesthesia maintenance with sevoflurane-only, then will be switched after 30 minutes to anesthesia with propofol-only.
  Interventions: Drug: Propofol 10 MG/ML
- Group B (Experimental): Group B will begin anesthesia with propofol-only then will be switched to sevoflurane-only.
  Interventions: Drug: Sevoflurane Inhalant Product

INTERVENTIONS:
Drug: Sevoflurane Inhalant Product — This study will perform intra-operative sonographic ONSD measurements in order to compare the change in ONSD during transition from inhalational maintenance anesthesia (using sevoflurane) to total intravenous anesthesia (TIVA) using propofol.
  Arms: Group B
Drug: Propofol 10 MG/ML — This study will perform intra-operative sonographic ONSD measurements in order to compare the change in ONSD during transition from inhalational maintenance anesthesia (using sevoflurane) to total intravenous anesthesia (TIVA) using propofol.
  Arms: Group A

SUMMARY:
We will prospectively compare change in ONSD during anesthesia with sevoflurane-only versus anesthesia with propofol-only in two groups of patients undergoing urologic and gynecologic surgery in the steep Trendelenburg position. We hypothesize that there will be a significant decrease in the size of ONSD during transition from sevoflurane-only anesthesia to propofol-only anesthesia.

DETAILED DESCRIPTION:
Steep Trendelenburg positioning is required for optimal surgical exposure for certain procedures, including robotic assisted laparoscopic urologic and gynecologic procedures. The position is associated with increased intracranial pressure (ICP) and its complications such as post-operative vision loss (POVL) and post-op delirium [Lee 2013]. Therefore, it is essential to measure ICP intra-operatively in order to implement real time management. The gold standard for ICP measurement is an external ventricular drain (EVD). However, it is invasive and not practical for the majority of non-neurosurgical procedures. Trans-ocular ultrasound measurement of Optic nerve sheath diameter (ONSD) is a non-invasive alternative for ICP measurement [Tayal et al 2007; Nash et al 2016]. Compared to EVD it is non-invasive, less expensive and efficient. It has been validated as a screening tool for identification of patients with elevated ICP who required treatment in several larger studies [Nash et al 2016; Blecha et al 2017]. During these procedures prior pre-cautions to prevent increased ICP focused on fluid restriction/selection. Ultrasound measurement of ONSD has not been routinely employed. Furthermore, consideration has rarely been given to the benefits of total intravenous anesthesia (TIVA) rather than volatile anesthetics for anesthesia maintenance during these procedures. Considering the complications of increased ICP, sonographic measurement could prove to be a practical method to efficiently monitor the ICP surrogate [Riaz et al 2016; Nash et al 2016; Banerjee et al 2017]. This study will perform intra-operative sonographic ONSD measurements in order to compare the change in ONSD during transition from inhalational maintenance anesthesia (using sevoflurane) to total intravenous anesthesia (TIVA) using propofol.

While other studies have demonstrated that the use of pneumoperitoneum and steep Trendelenburg positioning can lead to an increase in ICP as determined by use of ONSD (Robba et al. 2016), this study describes the added role of ONSD measurement for guiding the choice of anesthesia maintenance (TIVA vs sevoflurane) during surgery in the steep-Trendelenburg position.

ELIGIBILITY:
Inclusion Criteria:

All patients scheduled to undergo surgery in the steep Trendelenburg position at SUNY Downstate Medical Center.

Exclusion Criteria:

< 18 years old Pregnancy Pre-existing eye disease Prior ophthalmic surgery Inability to tolerate steep Trendelenburg position Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-01-17 (Estimated); Study Completion 2022-01-17 (Estimated)

PRIMARY OUTCOMES:
Sevoflurane Versus Propofol on Optic Nerve Sheath Diameter During Anesthesia in Steep Trendelenburg Position | 2 years
  1. Percentage of change in ONSD during anesthesia with sevoflurane-only versus propofol-only in two groups of patients undergoing urologic and gynecologic surgery in the steep Trendelenburg position.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee LA. Perioperative visual loss and anesthetic management. Curr Opin Anaesthesiol. 2013 Jun;26(3):375-81. doi: 10.1097/ACO.0b013e328360dcd9. PMID 23614957
- [Background] Moretti R, Pizzi B. Ultrasonography of the optic nerve in neurocritically ill patients. Acta Anaesthesiol Scand. 2011 Jul;55(6):644-52. doi: 10.1111/j.1399-6576.2011.02432.x. Epub 2011 Apr 4. PMID 21463263
- [Background] Blecha S, Harth M, Schlachetzki F, Zeman F, Blecha C, Flora P, Burger M, Denzinger S, Graf BM, Helbig H, Pawlik MT. Changes in intraocular pressure and optic nerve sheath diameter in patients undergoing robotic-assisted laparoscopic prostatectomy in steep 45 degrees Trendelenburg position. BMC Anesthesiol. 2017 Mar 11;17(1):40. doi: 10.1186/s12871-017-0333-3. PMID 28284189
- [Background] Tranquart F, Berges O, Koskas P, Arsene S, Rossazza C, Pisella PJ, Pourcelot L. Color Doppler imaging of orbital vessels: personal experience and literature review. J Clin Ultrasound. 2003 Jun;31(5):258-73. doi: 10.1002/jcu.10169. PMID 12767021
- [Background] Riaz R, Khuba S, Shamim R, Patro A. Ultrasonographic optic nerve sheath diameter measurement in overweight parturient with intracranial tumour: Guiding choice of anaesthesia. Indian J Anaesth. 2016 Oct;60(10):775-777. doi: 10.4103/0019-5049.191701. No abstract available. PMID 27761045
- [Background] Banerjee A, Bala R, Saini S. Ultrasonographic measurement of optic nerve sheath diameter: A point of care test helps in prognostication of Intensive Care Unit patients. Indian J Anaesth. 2017 Mar;61(3):262-265. doi: 10.4103/ija.IJA_473_16. PMID 28405042
- [Background] Tayal VS, Neulander M, Norton HJ, Foster T, Saunders T, Blaivas M. Emergency department sonographic measurement of optic nerve sheath diameter to detect findings of increased intracranial pressure in adult head injury patients. Ann Emerg Med. 2007 Apr;49(4):508-14. doi: 10.1016/j.annemergmed.2006.06.040. Epub 2006 Sep 25. PMID 16997419
- [Background] Kim JY, Min HG, Ha SI, Jeong HW, Seo H, Kim JU. Dynamic optic nerve sheath diameter responses to short-term hyperventilation measured with sonography in patients under general anesthesia. Korean J Anesthesiol. 2014 Oct;67(4):240-5. doi: 10.4097/kjae.2014.67.4.240. Epub 2014 Oct 27. PMID 25368781
- [Background] Robba C, Cardim D, Donnelly J, Bertuccio A, Bacigaluppi S, Bragazzi N, Cabella B, Liu X, Matta B, Lattuada M, Czosnyka M. Effects of pneumoperitoneum and Trendelenburg position on intracranial pressure assessed using different non-invasive methods. Br J Anaesth. 2016 Dec;117(6):783-791. doi: 10.1093/bja/aew356. PMID 27956677